CLINICAL TRIAL: NCT01535027
Title: Phase IV Study Teriparatide and Antiresorptive Combination Treatment Subsequent to 9 Months of Teriparatide Monotherapy
Brief Title: Combined Administration of Teripapartide and Antiresorptive Agents in Postmenopausal Osteoporosis
Acronym: Confors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christian Muschitz, Principle Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vinforce-003
Record Dates: First submitted 2011-12-20; First posted 2012-02-17 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Osteoporosis
Keywords: teriparatide; alendronate; raloxifene; bone mineral density
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Raloxifene Hydrochloride; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Teriparatide (Active Comparator): 18 months of daily 20 ug sc. teriparatide monotherapy (TPTD)
  Interventions: Drug: teriparatide
- Teriparatide and Raloxifene (Active Comparator): 9 months teriparatide 20 ug/day sc. monotherapy (TPTD) continued by combination therapy of raloxifene 60 mg/day orally(RAL)and TPTD for another 9 months
  Interventions: Drug: teriparatide and raloxifene
- Teriparatide and Alendronate (Active Comparator): 9 months teriparatide monotherapy 20 ug/day sc.(TPTD) continued by combination therapy of alendronate 70 mg/week orally(ALN)and TPTD for another 9 months
  Interventions: Drug: teriparatide and alendronate

INTERVENTIONS:
Drug: teriparatide — teriparatide 20 ug/day, sc.
  Other Names: Forteo
  Arms: Teriparatide
Drug: teriparatide and raloxifene — teriparatide 20 ug/day sc. raloxifene 60mg oral daily
  Other Names: Forteo; Evista
  Arms: Teriparatide and Raloxifene
Drug: teriparatide and alendronate — teriparatide 20 ug/day sc. alendronate 70mg oral weekly
  Other Names: Forteo; Fosamax
  Arms: Teriparatide and Alendronate

SUMMARY:
Increased bone formation in the absence of accelerated resorption is resulting in a marked anabolic response to teriparatide (TPTD) during the early phase after treatment initiation. Months later, due to coupling mechanism, the sustained increase of bone formation and ongoing anabolic effects are accompanied by significantly increased bone resorption as well. Antiresorptives influence the balance of bone formation and resorption. Therefore the investigators aim is to investigate the effects of the addition of antiresorptives to the second half of TPTD cycle when resorption is already also markedly elevated.

DETAILED DESCRIPTION:
We prospectively randomize 125 postmenopausal women after 9 months of TPTD treatment into three different open-label groups for another 9 months: either alendronate (ALN, 70 mg/week), raloxifene (RAL, 60 mg/day) or no medication (TPTD mono) on top of ongoing TPTD treatment.

All subjects receive daily supplementation of 1000mg calcium and 800 IU vitamin D.

Serum level of intact amino terminal propeptide of type I procollagen (PINP) and type 1 collagen cross-linked C-telopeptide (CTX) as well as DXA measurement at the spine, total hip and femoral neck BMD are evaluated at TPTD treatment initiation, at baseline of randomization to antiresorptive therapy as well as at 3 and 9 months during the combination treatment.Volumetric BMD values will be also determined.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory postmenopausal women at least 55 years of age
* Patients with "unsatisfactory clinical response to previous antiresorptive therapy" according to the national reimbursement criteria of Austria (either new clinical or radiographic fragility fracture on ≥ 2 years and/or accelerated bone loss of ≥ 3.5%/year on antiresorptive treatment; discontinuation of oral antiresorptive treatment due to side-effects and substantial risk for osteoporotic fracture defined by a T-Score ≤ -2.5 or ≥ 2 clinical risk factors according to the FRAX™-algorithm)and consequently started with teriparatide treatment
* Patients treated with teriparatide (20 ug/day) currently and since 9 months for postmenopausal osteoporosis
* Lumbar spine, femoral neck, and total hip evaluable by dual energy x ray absorptiometry (DXA)
* Normal or clinically non-significant abnormal laboratory values (as defined by the investigator)
* Without language barrier, cooperative, expected to return for all follow-up procedures, and who give informed consent before entering the study and after being informed of the medications and procedures to be used in this study

Exclusion Criteria:

* History of bone metabolic diseases, Paget's disease, renal osteodystrophy, osteomalacia, any secondary causes of osteoporosis, hyperparathyroidism (uncorrected), and intestinal malabsorption
* History of malignant neoplasms in the prior 5 years, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. If malignant neoplasm was ever diagnosed, patient must presently be free of disease
* History of nephrolithiasis or urolithiasis in the prior 2 years. Patients with any documented history of nephro- or uro-lithiasis must have had an appropriate imaging procedure within the prior 6 months, such as, an intravenous pyleogram (IVP), supine radiograph of the kidney ureter bladder, or renal ultrasound, which must document the absence of stones
* Abnormal thyroid function at any time in the prior 6 months. Patients with chronic hypothyreosis and adequate substitution therapy are permitted
* Active liver disease (liver enzymes more than three times the upper limit of normal) or clinical jaundice
* Significantly impaired renal function. This is defined as serum creatinine >1.8 mg/dL
* Treatment with bone active agent other than teriparatide in the prior 9 months

Ages: 55 Years to 88 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Differences in changes of areal lumbar spine BMD between the three treatment groups | Evaluation after 9, 12 and 18 months of TPTD
  Primary objective To investigate the changes in lumbar spine BMD of patients among the three treatment groups

SECONDARY OUTCOMES:
Differences in changes of BMDs and markers of bone turnover among the three treatment groups after 18 months TPTD treatment | Evaluation after 9, 12 and 18 months of TPTD treatment
  Secondary objectives
  * Differences in change of biochemical markers of bone turnover (serum CTX and serum PINP) between treatment groups
  * Differences in change of the additional DXA results in the hip scan (neck, upper neck, nape, Wards, Troch, shaft, total hip [g/cm²]) of patients between treatment groups
  * To investigate the volumetric changes of vertebral and hip BMD by quantitative computertomography of patients between treatment groups
  * To investigate safety and tolerability of the treatments

CONTACTS AND LOCATIONS:
Overall Officials: Christian Muschitz, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Muschitz C, Kocijan R, Fahrleitner-Pammer A, Pavo I, Haschka J, Schima W, Kapiotis S, Resch H. Overlapping and continued alendronate or raloxifene administration in patients on teriparatide: effects on areal and volumetric bone mineral density--the CONFORS Study. J Bone Miner Res. 2014 Aug;29(8):1777-85. doi: 10.1002/jbmr.2216. PMID 24619763
- See also: Homepage of Medical Department II, Vienna (German) — http://www.bhs-wien.at/index_html?sc=10355